CLINICAL TRIAL: NCT02562014
Title: Effect of Inulin and Resistant Starch on Postprandial Short Chain Fatty Acid, Glucose, Insulin and Gut Hormone Responses in Lean and Overweight Subjects.
Brief Title: Role of Colonic Short Chain Fatty Acids in Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Thomas Wolever, Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Protocol #27112
Record Dates: First submitted 2015-09-25; First posted 2015-09-29 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Glucose; Inulin; Resistant Starch

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lean (Other): Participants with body mass index <=25
  Interventions: Other: Glucose; Other: Inulin; Other: Resistant Starch
- Overweight (Other): Participants with body mass index >25
  Interventions: Other: Glucose; Other: Inulin; Other: Resistant Starch

INTERVENTIONS:
Other: Glucose — 75g glucose
Other: Inulin — 75g glucose plus 24g inulin
Other: Resistant Starch — 75g glucose plus 28.2g resistant starch

SUMMARY:
The excess production of colonic short-chain-fatty-acids (SCFA) has been implicated in the promotion of obesity, but colonic fermentation of dietary-fiber to SCFA may also play a role in preventing diabetes. The investigators aimed to compare the effects of two fermentable fibers (inulin and resistant-starch) on postprandial SCFA, glucose, insulin, free-fatty acids (FFA) and gut hormone responses and to compare the responses in healthy overweight and obese (OWO) vs lean (LN) participants. Methods: Using a randomized, single blind, crossover design, 13 OWO and 12 LN overnight fasted participants were studied on 3 separate occasions. On each day they consumed a 300 mL drink containing 75g glucose (Control) or 75g glucose plus 24g inulin (IN), or 28.2g resistant-starch (RS). A standard lunch was served 4 h after the test drink.

ELIGIBILITY:
Inclusion Criteria:

* non-pregnant
* body mass index >=20 and <=35

Exclusion Criteria:

* history of diabetes mellitus
* history of cardiovascular disease
* history of bowel disease
* history of kidney disease
* history of liver disease
* use of antibiotics within 3 months of enrolment
* unusual dietary habits
* fasting glucose >6.9mmol/L
* hematocrit below normal range for age and sex

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-02; Primary Completion 2012-07 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Incremental area under the serum acetate response curve | For 6 hours after consuming the test meal

SECONDARY OUTCOMES:
Incremental area under the serum propionate response curve | For 6 hours after consuming the test meal
Incremental area under the serum butyrate response curve | For 6 hours after consuming the test meal
Incremental area under the breath hydrogen response curve | For 6 hours after consuming the test meal
Incremental area under the breath methane response curve | For 6 hours after consuming the test meal
Incremental area under the serum glucose response curve | For 4 hours after consuming the test meal
Incremental area under the serum glucose response curve | For 2 hours after consuming the standard lunch
Incremental area under the serum insulin response curve | For 4 hours after consuming the test meal
Incremental area under the serum insulin response curve | For 2 hours after consuming the standard lunch
Incremental area under the serum c-peptide response curve | For 4 hours after consuming the test meal
Incremental area under the serum c-peptide response curve | For 2 hours after consuming the standard lunch
Total area under the serum free-fatty acid response curve | For 4 hours after consuming the test meal
Total area under the serum free-fatty acid response curve | For 2 hours after consuming the standard lunch

OTHER OUTCOMES:
Incremental area under the serum glucagon-like peptide-1 response curve | For 4 hours after consuming the test meal
Incremental area under the serum glucagon-like peptide-1 response curve | For 2 hours after consuming the standard lunch
Incremental area under the serum peptide-YY response curve | For 4 hours after consuming the test meal
Incremental area under the serum peptide-YY response curve | For 2 hours after consuming the standard lunch
Incremental area under the serum ghrelin response curve | For 4 hours after consuming the test meal
Incremental area under the serum ghrelin response curve | For 2 hours after consuming the standard lunch

CONTACTS AND LOCATIONS:
Overall Officials: Thomas MS Wolever, MD, PhD, Principal Investigator — University of Toronto

REFERENCES:
- [Derived] Rahat-Rozenbloom S, Fernandes J, Cheng J, Wolever TMS. Acute increases in serum colonic short-chain fatty acids elicited by inulin do not increase GLP-1 or PYY responses but may reduce ghrelin in lean and overweight humans. Eur J Clin Nutr. 2017 Aug;71(8):953-958. doi: 10.1038/ejcn.2016.249. Epub 2016 Dec 14. PMID 27966574
- [Derived] Rahat-Rozenbloom S, Fernandes J, Cheng J, Gloor GB, Wolever TM. The acute effects of inulin and resistant starch on postprandial serum short-chain fatty acids and second-meal glycemic response in lean and overweight humans. Eur J Clin Nutr. 2017 Feb;71(2):227-233. doi: 10.1038/ejcn.2016.248. Epub 2016 Dec 14. PMID 27966565